CLINICAL TRIAL: NCT04525027
Title: Predictive Ability of Intra-Abdominal Pressure for Mortality in Patients With Severe Acute Pancreatitis: A Prospective Observational Study
Brief Title: Predictive Ability of Intra-Abdominal Pressure for Mortality in Patients With Severe Acute Pancreatitis
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, VAMSIDHAR, Trainee, Sir Ganga Ram Hospital
Other Study IDs: EC/12/19/1650
Record Dates: First submitted 2020-08-18; First posted 2020-08-24 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Acute Pancreatitis; Intra-Abdominal Hypertension
Keywords: severe acute pancreatitis; intra abdominal pressure; mortality; intra abdominal hypertension
MeSH Terms: conditions — Pancreatitis; Intra-Abdominal Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (2):
- survivors
  Interventions: Diagnostic Test: intra-abdominal pressure in severe acute pancreatitis
- non survivors
  Interventions: Diagnostic Test: intra-abdominal pressure in severe acute pancreatitis

INTERVENTIONS:
Diagnostic Test: intra-abdominal pressure in severe acute pancreatitis — daily intra abdominal pressures in patients admitted to ICU will be measured and noted for intial 5 days and followed up until end outcome

SUMMARY:
Severe Acute Pancreatitis (SAP) is an acute inflammatory condition of the pancreas characterized by organ dysfunction and increased mortality. Increased Intra-abdominal Pressure(IAP) in SAP is a result of inflammation of pancreatic and peripancreatic tissue, aggressive fluid resuscitation and increased capillary permeability, which is associated with organ dysfunction, by limiting the vascular supply to the tissue. Abdominal Compartment Syndrome (ACS) is defined as IAP greater than 20 mm of Hg and is considered an abdominal catastrophe. Intra-abdominal Hypertension (IAH, Intra-abdominal pressure > 12mm of Hg), may contribute to early organ dysfunction, ACS and eventually hemodynamic collapse if left untreated. This signifies the need for determining the burden of the condition and identifying the high risk patient group who are prone to develop IAH /ACS and predicting mortality associated with the condition. Measurement of IAP will be done indirectly by measuring intravesicular pressure using modified kron's method. IAP will be measured at the time of admission into Intensive Care Unit (ICU) and every day thereafter during the initial five days of ICU admission. Any reading of IAP ≥12 mm of Hg shall be considered as IAH. SOFA and APACHE II score will be noted on the day of admission in the ICU. Any interventions, surgical or non surgical as per clinician's decision will be recorded. The patients will be followed up until discharge or mortality until 30 days. The proposed study aims to assess the predictive ability of IAP during the first 5 days of ICU admission for predicting mortality in patients with SAP. Prediction accuracy will also be compared with SOFA and APACHE II scores.

ELIGIBILITY:
Inclusion Criteria:

>Patients with severe acute pancreatitis in the age group of 18-65 years admitted to ICU within 72 hours of onset of symptoms

Exclusion Criteria:

* Previous history of any abdominal or pelvic surgery
* Known case of bladder tumor or bladder abnormality.
* Difficulty in urinary catheterization
* Use of neuromuscular blockade
* Pregnant patients

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients of acute severe pancreatitis admitted to ICU within 72 hours of symptom onset
Sampling Method: Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2019-12-26 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days from inclusion date

CONTACTS AND LOCATIONS:
Overall Officials: vinod singh, MD, Study Chair — Sir Ganga Ram Hospital
Locations (1):
- Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided